CLINICAL TRIAL: NCT02182856
Title: A Randomised, Double-blind, Active-controlled, Within-patient Trial Comparing the Effect of Single Doses of Nebulised Ipratropium 500µg, Salbutamol Sulphate 3mg, Salbutamol 6mg and the Combination Therapy Salbutamol Sulphate 3 mg Plus Ipratropium 500µg on Arterial Oxygen Saturation in Patients With Stable, Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Ipratropium or Salbutamol Sulphate Alone or Combination Therapy Salbutamol and Ipratropium in Patients With COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.39
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Ipratropium bromide/salbutamol sulphate (Experimental): Randomised sequence of four different treatments
  1. Ipratropium bromide 500 µg/salbutamol sulphate 3 mg
  2. Ipratropium 500 µg
  3. Salbutamol sulphate 3 mg
  4. Salbutamol sulphate 6 mg
  Interventions: Drug: Ipratropium bromide 500 µg/salbutamol sulphate 3 mg; Drug: Ipratropium 500 µg; Drug: Salbutamol sulphate 3 mg; Drug: Salbutamol sulphate 6 mg

INTERVENTIONS:
Drug: Ipratropium bromide 500 µg/salbutamol sulphate 3 mg
  Other Names: Combivent® UDVs®
Drug: Ipratropium 500 µg
Drug: Salbutamol sulphate 3 mg
Drug: Salbutamol sulphate 6 mg

SUMMARY:
Study to compare the effects of nebulised salbutamol or ipratropium alone in patients with COPD with those of combined salbutamol and ipratropium nebuliser solution on arterial oxygen saturation (SaO2) and to characterise patients with COPD (chronic obstructive pulmonary disease) at risk of significant arterial oxygen desaturation following nebulised salbutamol.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with moderate to severe stable COPD:

  * Patients with a diagnosis of chronic bronchitis and/or emphysema
  * FEV1 <65% of predicted value without regard to prior treatment
  * Forced expiratory ration (FER = FEV1/VC) <70% of predicted value without regard to prior treatment
  * Patients must not have had a respiratory infection or an exacerbation of COPD during the four weeks immediately prior to entering the trial
  * Patients must not have changed their normal treatment for COPD during the four weeks immediately prior to entering the trial
* Patient aged ≥40 years
* Patients with a smoking history of ≥15 pack-years
* Patients must have given informed consent to participate in the trial

Exclusion Criteria:

* Patients with a diagnosis of asthma, bronchiectasis, cystic fibrosis or bronchiolitis obliterans
* Patients with any of the following:

  * untreated angle closure glaucoma
  * hypertrophic obstructive cardiomyopathy
  * tachyarrhythmia
  * recent myocardial infarction (within six months of screening visit)
  * severe organic cardiac or vascular disorder
  * untreated hyperthyroidism
  * diabetes mellitus (after approval of Protocol Amendment 1, the inclusion of well controlled diabetic patients was allowed)
* Patients who are pregnant, or who are planning a pregnancy, and nursing mothers
* Patients known to be hypersensitive to anticholinergic drugs or to β2 agonists
* Patients known to abuse drugs or alcohol
* Patients, who in the opinion of the investigator, are likely not to co-operate with any of the requirements of the trial
* Patients with a PaO2 (arterial carbon dioxide tension) <56 mmHg (7.5 kPa) at rest while breathing air without regard to prior treatment
* Patients with a SaO2 ≤85% at rest while breathing air without regard to prior treatment
* Patients who are taking part in another investigation, and patients who have participated in another clinical trial during the three months immediately preceding entry to this trial
* Patients on home oxygen concentrator therapy
* Patients who have previously participated in the randomised phase of this trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1998-02; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve of arterial oxygen saturation (SaO2) | over 70 min observation period from each start of nebulisation

SECONDARY OUTCOMES:
Forced expiratory volume in the first second of expiration (FEV1) | up to 60 min after end of nebulisation
Relaxed (expiratory) vital capacity (VC) | up to 60 min after end of nebulisation
Forced (expiratory) vital capacity (FVC) | up to 60 min after end of nebulisation
Forced expiratory ratio (FER) | up to 60 min after end of nebulisation